CLINICAL TRIAL: NCT04261400
Title: MAMAACT Intervention for Improved Reproductive Health - a Feasibility Study
Brief Title: Early Evaluation of the MAMAACT Trial
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: University of Copenhagen (Other)
Collaborators: Hvidovre University Hospital (Other); The Danish Council for Strategic Research (Other)
Responsible Party: Principal Investigator, Sarah Fredsted Villadsen, Assistant Professor / Ph.D, University of Copenhagen
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: MAMAACT#1
Record Dates: First submitted 2020-02-04; First posted 2020-02-07 (Actual); Last update posted 2020-02-07 (Actual); Status verified 2020-02

CONDITIONS: Pregnancy Complications
MeSH Terms: conditions — Pregnancy Complications

STUDY DESIGN:
Intervention Model Description: The intervention package was provided to midwives working at two specific antenatal care facilities and the women attending care at these facilities received the health education material.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- MAMAACT (Experimental): Post graduate training of midwives in intercultural communication and health education materials for the pregnant women.
  Interventions: Behavioral: MAMAACT
- Control (No Intervention): Care as usual

INTERVENTIONS:
Behavioral: MAMAACT — Improved communication regarding warning signs of pregnancy complications
  Arms: MAMAACT

SUMMARY:
The MAMAACT#1 project's aim was to reduce ethnic disparity in stillbirth and infant death by improving the management of pregnancy complications through timely and appropriate response to warning signs of pregnancy. The intervention consisted of a training program for midwives and health education materials for pregnant women. The aim of the feasibility trial was to analyze the acceptability and feasibility of the MAMAACT intervention using mini-group interviews with midwives and to pilot outcome evaluation using surveys.

DETAILED DESCRIPTION:
The MAMAACT project's aim was to reduce ethnic disparity in stillbirth and infant death by improving the management of pregnancy complications through timely and appropriate response to warning signs of pregnancy. The intervention was co-created with midwives at Hvidovre Hospital, the largest maternity ward in Denmark. The intervention consisted of a 5-hour training session for midwives in intercultural communication followed by three dialogue meetings in smaller groups. The first midwife visit was extended with 5 minutes allowing for more communication and health education on body symptoms. The women were given a leaflet and a mobile application at this first visit that were describing when and how to respond to warning signs during pregnancy. Both the leaflet and application were available in Danish, Arabic, Persian, English, Somali, Turkish, and Urdu.

The intervention was a complex intervention, and this phase was a feasibility study preceding a national trial. This feasibility trial was tested at one hospital 2014-2015. The national trial 2017-2021 is registered with ClinicalTrials.gov Identifier: NCT03751774.

The hospital had four antenatal clinics and the intervention was implemented at two clinics, while two served as control clinics. The MAMAACT leaflet and app were distributed to all pregnant women at the two intervention clinics, equivalent n=2000, attending antenatal care during the test period.

The aim of the feasibility trial was to analyze the acceptability and feasibility of the trial and to pilot outcome evaluation using surveys in a difference in difference design. The acceptability and feasibility of the intervention were evaluated using mini-groups interviews with midwives in the intervention arm. The difference in difference study was piloted comparing change in outcomes of women from the intervention arm from before the intervention to after the intervention relative to the change in the control arm. Survey assessed outcomes were women's' knowledge about warning signs of pregnancy complications, health system navigation and satisfaction with the midwifery based antenatal care.

ELIGIBILITY:
Inclusion Criteria:

* Pregnant in gestational week 27+0-31+6 , affiliated to Hvidovre hospital, seen for antenatal care during recruitment weeks.

Exclusion Criteria:

* Not speaking Danish, English, Urdu, Turkish, Somali, Persian or Arabic.

Ages: 13 Years to 50 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult
Gender Based: Yes — Pregnant women
Enrollment: 2000 (Actual)
Dates: Start 2014-01-01 (Actual); Primary Completion 2015-06-01 (Actual); Study Completion 2015-06-01 (Actual)

PRIMARY OUTCOMES:
Womens satisfaction with midwifery based antenatal care | Assessed among women in pregnancy week 27+0 to 31+6
  Changed level of satisfaction with midwifery based antenatal care among pregnant women. Satisfaction was measured by the question: "I was satisfied with the conversation that I had with the midwife" with four response categories: Strongly agree, Agree, Disagree, or Strongly disagree. This item was an adapted version of the item from the Maternity study in Jimma, Ethiopia (Villadsen, S.F., Negussie, D., GebreMariam, A. et al. Antenatal care strengthening for improved quality of care in Jimma, Ethiopia: an effectiveness study. BMC Public Health 15, 360 (2015). https://doi.org/10.1186/s12889-015-1708-3).

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Johnsen H, Ghavami Kivi N, Morrison CH, Juhl M, Christensen U, Villadsen SF. Addressing ethnic disparity in antenatal care: a qualitative evaluation of midwives' experiences with the MAMAACT intervention. BMC Pregnancy Childbirth. 2020 Feb 19;20(1):118. doi: 10.1186/s12884-020-2807-4. PMID 32075593